CLINICAL TRIAL: NCT06263231
Title: A Multicenter, Randomized, Phase 3 Study to Assess the Efficacy and Safety of INtratumorally Administered INT230-6 (SHAO, VINblastine, CIsplatin) Compared With US Standard of Care in Adults With Locally Recurrent, InoperaBLE, or Metastatic Soft Tissue Sarcomas (INVINCIBLE-3)
Brief Title: A Study to Investigate Efficacy & Safety of Intratumoral INT230-6 Compared to US Standard of Care in Adults With Soft Tissue Sarcomas (INVINCIBLE-3)
Acronym: INVINCIBLE-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intensity Therapeutics, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IT-03
Record Dates: First submitted 2024-02-01; First posted 2024-02-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — eribulin; Trabectedin; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- INT230-6 Monotherapy (Experimental): INT230-6 administered intratumorally. Participants will be dosed every 2 weeks (± 2 days) for up to a total of 5 treatment sessions (e.g., Days 1, 15, 29, 43 and 57). Once the participant has completed the treatment phase, they will continue into a 22-month maintenance phase, where investigators may inject new lesions or previously injected lesions with up to 175 mL of INT230-6 every 12 weeks (Q12W) ± 14 days. Dose volume in a session is dependent on the participants presenting tumor burden.
  Interventions: Drug: INT230-6
- US Standard of Care (Active Comparator): Participants in this arm may receive any of the following depending on soft tissue sarcoma (STS) subtype and PI preference:
  * Pazopanib: 800 mg PO every day until clinical deterioration or disease progression
  * Trabectedin: 1.5 mg/m2 body surface area as 24-hour IV infusion every 3 weeks until clinical deterioration or disease progression
  * Eribulin:
  Non- European Union (EU) sites: 1.4 mg/m2 eribulin mesylate body surface area IV on Days 1 and 8 every 3 weeks until clinical deterioration or disease progression EU sites: 1.23 mg/m2 (free base) body surface area IV on Days 1 and 8 every 3 weeks until clinical deterioration or disease progression
  Interventions: Drug: Eribulin; Drug: Trabectedin; Drug: Pazopanib

INTERVENTIONS:
Drug: INT230-6 — INT230-6 is a fixed combination of cisplatin, vinblastine and SHAO.
  Arms: INT230-6 Monotherapy
Drug: Eribulin — Eribulin IV
  Arms: US Standard of Care
Drug: Trabectedin — Trabectedin infusion
  Arms: US Standard of Care
Drug: Pazopanib — Pazopanib pill
  Arms: US Standard of Care

SUMMARY:
To compare Overall Survival (OS) for INT230-6 vs United States (US) Standard of Care (SOC) in participants with unresectable or metastatic liposarcoma, undifferentiated pleomorphic sarcoma or leiomyosarcoma who have disease progression prior to study enrollment following no more than 2 standard therapies, which must have included an anthracycline-based regimen, unless contraindicated, and then a maximum of 1 additional regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is of any sex and must be ≥ 18 years old and provide written informed consent to participate in the study.

   Type of Participant and Disease Characteristics
2. Histologically proven, unresectable, locally advanced, or metastatic Soft Tissue Sarcoma (STS) only of the following subtypes: liposarcoma (dedifferentiated, myxoid, round cell or pleomorphic), leiomyosarcoma, and undifferentiated pleomorphic sarcoma. Participant must have a pathology report indicating the diagnosis of their STS.
3. Participant must have received at least 1 line of therapy for a STS and must have progressed following anthracycline-based or alternative standard therapies, except if medically contraindicated or refused by participant. Participant cannot have received more than 2 prior regiments for unresectable, locally advanced or metastatic STS.
4. Participant must have measurable disease per RECIST 1.1 criteria.
5. Participant must have at least 1 target tumor suitable for injection using routine image guidance ≥ 2 cm measurable by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI).
6. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 (see Section 11.7).
7. Participant must have adequate organ function as defined by screening laboratory values that must meet the following criteria:

   1. Neutrophils ≥ 1500/μL (≥ 1.5× 109/L).
   2. Prothrombin Time (PT), and International Normalized Ratio (INR) ≤ 1.5× Upper Limit of Normal (ULN), platelets ≥ 100,000/μL (≥ 10× 109/L); hemoglobin ≥ 9 g/dL. Criteria must be met without erythropoietin dependency and without packed red blood cell transfusion within the last 2 weeks.
   3. Creatinine within normal range; or calculated creatinine clearance > 50 mL/min by the Cockcroft-Gault equation.
   4. Alanine Aminotransferase (ALT) Serum Glutamic-Oxaloacetic Transaminase (SGOT)/ Aspartate Aminotransferase (AST) Serum Glutamic-Pyruvic Transaminase (SGPT) ≤ 2.5× ULN without, and ≤ 5× ULN with hepatic metastases.
   5. Bilirubin ≤ 1.5× ULN (except participants with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL [< 52 µmol/L]).
   6. Creatine phosphokinase < 2.5× ULN Sex and Contraceptive/Barrier Requirements
8. A female participant is eligible to participate if she is not pregnant (as demonstrated by pregnancy testing prior to each treatment; performed at least monthly), not breastfeeding, and at least 1 of the following conditions applies:

   1. Not a Woman of Childbearing Potential (WOCBP). Women of non-childbearing potential are defined as women with functioning ovaries with a documented history of tubal ligation or hysterectomy or females who are post menopausal, as defined by 12 months of spontaneous amenorrhea with an appropriate clinical profile, e.g., age appropriate, > 45 years, in the absence of hormone replacement therapy. In questionable cases, a blood sample for Follicle Stimulating Hormone (FSH) and estradiol will be obtained to confirm childbearing potential.
   2. A WOCBP who may become pregnant or who is sexually active with a partner and who could become pregnant agrees to use a highly effective form of contraception during the study and for at least 7 months after the end of study intervention (see Section 11.5.2 for highly effective methods of contraception).
9. Male participants with female partners of childbearing potential must agree to use contraception and refrain from sperm donation during the study and for 6 months after the end of study intervention (Section 11.5.2.2).

Exclusion Criteria:

Informed Consent:

1. Adult participants who lack capacity to consent without a legally authorized representative will be excluded from this study.

   Medical Conditions:
2. Prior primary or metastatic brain or meningeal tumors unless clinically and radiographically stable as well as off-steroid therapy for at least 2 months.
3. History of severe hypersensitivity reactions to US SOC agents and vinblastine or cisplatin or other products of the same class and their excipients.
4. Histologically proven, unresectable, locally advanced or metastatic STS subtypes other than those specified, for example excluded subtypes include liposarcoma (well differentiated), desmoid or dermatofibrosarcoma protuberans.
5. Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or superficial bladder cancer, or any other cancer from which the participant has been disease-free for at least 2 years.
6. Underlying medical condition that, in the investigator's opinion, will make the administration of study intervention hazardous or obscure the interpretation of toxicity determination or Adverse Events (AEs).
7. Concurrent medical condition requiring the use of immunosuppressive medications, or systemic corticosteroids (topical steroids are permitted); systemic corticosteroids must be discontinued at least 4 weeks prior to dosing.

   Inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if the participant is on a stable dose. Non-absorbed intra-articular steroid injections will be permitted. Use of steroids as prophylactic treatment for participants with contrast allergies to diagnostic imaging contrast dyes will be permitted.
8. Participants who require uninterrupted anticoagulants of any type or is on daily aspirin therapy or NSAIDS.
9. Known significant chronic liver disease, such as cirrhosis or active hepatitis (potential participants who test positive for hepatitis B surface antigen or hepatitis C antibodies are allowed provided they do not have active disease requiring antiviral therapy).
10. Myocardial infarction within 6 months before enrollment, New York Heart Association Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease or electrocardiographic evidence of acute ischemic or active conduction system abnormalities.
11. Uncontrolled intercurrent illness including, but not limited to, poorly controlled hypertension or diabetes, ongoing active infection or psychiatric illness/social situation that may potentially impair the participant's compliance with study procedures.
12. Participants with a Corrected QT interval (QTc) of >450 ms for men and >470 ms for women, or with a history of serum electrolyte abnormalities known to prolong the QT interval such hypocalcemia, hypokalemia, and hypomagnesemia, or a family or personal history of congenital long QT syndrome.
13. Participants actively receiving therapy with strong Cytochrome P450 3A4 isoenzyme (CYP3A4) inhibitors (e.g, erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil).
14. Participants actively receiving therapy with medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study intervention.

    Prior/Concomitant Therapy
15. Prior chemotherapy or immunotherapy (tumor vaccine, cytokine or growth factor given to control the cancer: systemic or IT) must have been completed at least 4 weeks prior to dosing (with the exception of kinase inhibitors or other short half-life drugs, a 2-week washout is acceptable prior to treatment) and all AEs have either returned to baseline or stabilized. Note: participants who have received prior platinum therapy are eligible irrespective of their response. If participant had received one of the 3 US SOC study regimens prior to enrollment, that previous US SOC cannot be assigned in this study.
16. Prior systemic radiation therapy (IV, intrahepatic or oral) completed at least 4 weeks prior to study intervention administration. Prior focal radiotherapy completed at least 2 weeks prior to study intervention administration.

    a. Prior major treatment-related surgery completed at least 4 weeks prior to study intervention administration.
17. Use of other investigational drugs (drugs not marketed for any indication) within 28 days prior to study intervention administration.
18. Received a live vaccine within 6 weeks of first dose of study intervention.
19. Received a Coronavirus Disease (COVID-19) vaccine less than 1 week prior to dosing (Cycle 1/Day 1) and/or during the study received a COVID-19 vaccine or booster less than 3 weeks ahead of a tumor assessment.

    Other Exclusion Criteria
20. Pregnancy Exclusion: A WOCBP who has a positive pregnancy test (e.g., within 72 hours) prior to treatment. If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of randomization until the documented date of death from any cause for a period of up to 2 years, unless superiority is demonstrated sooner or 80% of deaths during the study period.
  To compare OS for INT230-6 vs US Standard of Care (SOC) in participants with unresectable or metastatic liposarcoma, undifferentiated pleomorphic sarcoma or leiomyosarcoma who have disease progression prior to study enrollment following no more than 2 standard therapies, which must have included an anthracycline-based regimen, unless contraindicated, and then a maximum of 1 additional regimen.

SECONDARY OUTCOMES:
Overall Survival (OS) For INT230-6 Compared to OS for Standard of Care (SOC) for Participants with leiomyosarcoma | From date of randomization until the documented date of death from any cause for a period of up to 2 years, unless superiority is demonstrated sooner or 80% of deaths during the study period.
  To compare OS for INT230-6 vs US SOC in participants with leiomyosarcoma
Overall Survival (OS) For INT230-6 Compared to OS for Standard of Care (SOC) for Participants with liposarcoma | From date of randomization until the documented date of death from any cause for a period of up to 2 years, unless superiority is demonstrated sooner or 80% of deaths during the study period.
  To compare OS for INT230-6 vs US SOC in participants with liposarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Christian F. Meyer, MD, PhD, MS, Principal Investigator — Johns Hopkins University
Locations (17):
- United States (10):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of California Los Angeles (UCLA) - Santa Monica Cancer Care, Santa Monica, California
  - Yale School of Medicine - Smilow Cancer Hospital - Yale - New Haven Hospital Location, New Haven, Connecticut
  - Profound Research LLC, Farmington Hills, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Duke Cancer Center, Durham, North Carolina
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - University of Pennsylvania - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Temple University - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Centre Leon Berard, Lyon, France
- Germany (2):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Universitäres Krebszentrum (UCCL), Leipzig
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall Hebron, Barcelona
  - Centro Integral Oncologico Clara Campal (HM CIOCC), Madrid

IPD SHARING:
Plan to Share IPD: Yes
General Data Protection Regulation (GDPR) and HIPPA privacy laws will be followed for sharing of any data.
Supporting Information: Study Protocol, ICF
Time Frame: During the study for a period of 4 years.

REFERENCES:
- [Background] Billingsley KG, Burt ME, Jara E, Ginsberg RJ, Woodruff JM, Leung DH, Brennan MF. Pulmonary metastases from soft tissue sarcoma: analysis of patterns of diseases and postmetastasis survival. Ann Surg. 1999 May;229(5):602-10; discussion 610-2. doi: 10.1097/00000658-199905000-00002. PMID 10235518
- [Background] Beaver JA, Hazarika M, Mulkey F, Mushti S, Chen H, He K, Sridhara R, Goldberg KB, Chuk MK, Chi DC, Chang J, Barone A, Balasubramaniam S, Blumenthal GM, Keegan P, Pazdur R, Theoret MR. Patients with melanoma treated with an anti-PD-1 antibody beyond RECIST progression: a US Food and Drug Administration pooled analysis. Lancet Oncol. 2018 Feb;19(2):229-239. doi: 10.1016/S1470-2045(17)30846-X. Epub 2018 Jan 18. PMID 29361469
- [Background] Bender LH, Abbate F, Walters IB. Intratumoral Administration of a Novel Cytotoxic Formulation with Strong Tissue Dispersive Properties Regresses Tumor Growth and Elicits Systemic Adaptive Immunity in In Vivo Models. Int J Mol Sci. 2020 Jun 24;21(12):4493. doi: 10.3390/ijms21124493. PMID 32599852
- [Background] Bloom AC, Bender LH, Tiwary S, Pasquet L, Clark K, Jiang T, Xia Z, Morales-Kastresana A, Jones JC, Walters I, Terabe M, Berzofsky JA. Intratumorally delivered formulation, INT230-6, containing potent anticancer agents induces protective T cell immunity and memory. Oncoimmunology. 2019 Jul 16;8(10):e1625687. doi: 10.1080/2162402X.2019.1625687. eCollection 2019. PMID 31646070
- [Background] Cassier PA, Polivka V, Judson I, Soria JC, Penel N, Marsoni S, Verweij J, Schellens JH, Morales-Barrera R, Schoffski P, Voest EE, Gomez-Roca C, Evans TR, Plummer R, Gallerani E, Kaye SB, Olmos D. Outcome of patients with sarcoma and other mesenchymal tumours participating in phase I trials: a subset analysis of a European Phase I database. Ann Oncol. 2014 Jun;25(6):1222-8. doi: 10.1093/annonc/mdu108. Epub 2014 Mar 7. PMID 24608201
- [Background] Dasari S, Tchounwou PB. Cisplatin in cancer therapy: molecular mechanisms of action. Eur J Pharmacol. 2014 Oct 5;740:364-78. doi: 10.1016/j.ejphar.2014.07.025. Epub 2014 Jul 21. PMID 25058905
- [Background] Demetri GD, von Mehren M, Jones RL, Hensley ML, Schuetze SM, Staddon A, Milhem M, Elias A, Ganjoo K, Tawbi H, Van Tine BA, Spira A, Dean A, Khokhar NZ, Park YC, Knoblauch RE, Parekh TV, Maki RG, Patel SR. Efficacy and Safety of Trabectedin or Dacarbazine for Metastatic Liposarcoma or Leiomyosarcoma After Failure of Conventional Chemotherapy: Results of a Phase III Randomized Multicenter Clinical Trial. J Clin Oncol. 2016 Mar 10;34(8):786-93. doi: 10.1200/JCO.2015.62.4734. Epub 2015 Sep 14. PMID 26371143
- [Background] Gronchi A, Miah AB, Dei Tos AP, Abecassis N, Bajpai J, Bauer S, Biagini R, Bielack S, Blay JY, Bolle S, Bonvalot S, Boukovinas I, Bovee JVMG, Boye K, Brennan B, Brodowicz T, Buonadonna A, De Alava E, Del Muro XG, Dufresne A, Eriksson M, Fagioli F, Fedenko A, Ferraresi V, Ferrari A, Frezza AM, Gasperoni S, Gelderblom H, Gouin F, Grignani G, Haas R, Hassan AB, Hecker-Nolting S, Hindi N, Hohenberger P, Joensuu H, Jones RL, Jungels C, Jutte P, Kager L, Kasper B, Kawai A, Kopeckova K, Krakorova DA, Le Cesne A, Le Grange F, Legius E, Leithner A, Lopez-Pousa A, Martin-Broto J, Merimsky O, Messiou C, Mir O, Montemurro M, Morland B, Morosi C, Palmerini E, Pantaleo MA, Piana R, Piperno-Neumann S, Reichardt P, Rutkowski P, Safwat AA, Sangalli C, Sbaraglia M, Scheipl S, Schoffski P, Sleijfer S, Strauss D, Strauss S, Sundby Hall K, Trama A, Unk M, van de Sande MAJ, van der Graaf WTA, van Houdt WJ, Frebourg T, Casali PG, Stacchiotti S; ESMO Guidelines Committee, EURACAN and GENTURIS. Electronic address: clinicalguidelines@esmo.org. Soft tissue and visceral sarcomas: ESMO-EURACAN-GENTURIS Clinical Practice Guidelines for diagnosis, treatment and follow-up☆. Ann Oncol. 2021 Nov;32(11):1348-1365. doi: 10.1016/j.annonc.2021.07.006. Epub 2021 Jul 22. No abstract available. PMID 34303806
- [Background] Jones RL, Maki RG, Patel SR, Wang G, McGowan TA, Shalaby WS, Knoblauch RE, von Mehren M, Demetri GD. Safety and efficacy of trabectedin when administered in the inpatient versus outpatient setting: Clinical considerations for outpatient administration of trabectedin. Cancer. 2019 Dec 15;125(24):4435-4441. doi: 10.1002/cncr.32462. Epub 2019 Sep 10. PMID 31503332
- [Background] Lammers T, Peschke P, Kuhnlein R, Subr V, Ulbrich K, Huber P, Hennink W, Storm G. Effect of intratumoral injection on the biodistribution and the therapeutic potential of HPMA copolymer-based drug delivery systems. Neoplasia. 2006 Oct;8(10):788-95. doi: 10.1593/neo.06436. PMID 17032495
- [Background] Meyer M, Seetharam M. First-Line Therapy for Metastatic Soft Tissue Sarcoma. Curr Treat Options Oncol. 2019 Jan 24;20(1):6. doi: 10.1007/s11864-019-0606-9. PMID 30675651
- [Background] von Mehren M, Kane JM, Agulnik M, Bui MM, Carr-Ascher J, Choy E, Connelly M, Dry S, Ganjoo KN, Gonzalez RJ, Holder A, Homsi J, Keedy V, Kelly CM, Kim E, Liebner D, McCarter M, McGarry SV, Mesko NW, Meyer C, Pappo AS, Parkes AM, Petersen IA, Pollack SM, Poppe M, Riedel RF, Schuetze S, Shabason J, Sicklick JK, Spraker MB, Zimel M, Hang LE, Sundar H, Bergman MA. Soft Tissue Sarcoma, Version 2.2022, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2022 Jul;20(7):815-833. doi: 10.6004/jnccn.2022.0035. PMID 35830886
- [Background] Obeid M, Panaretakis T, Tesniere A, Joza N, Tufi R, Apetoh L, Ghiringhelli F, Zitvogel L, Kroemer G. Leveraging the immune system during chemotherapy: moving calreticulin to the cell surface converts apoptotic death from "silent" to immunogenic. Cancer Res. 2007 Sep 1;67(17):7941-4. doi: 10.1158/0008-5472.CAN-07-1622. PMID 17804698
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Padhani AR, Ollivier L. The RECIST (Response Evaluation Criteria in Solid Tumors) criteria: implications for diagnostic radiologists. Br J Radiol. 2001 Nov;74(887):983-6. doi: 10.1259/bjr.74.887.740983. No abstract available. PMID 11709461
- [Background] Phillips E, Jones RL, Huang P, Digklia A. Efficacy of Eribulin in Soft Tissue Sarcomas. Front Pharmacol. 2022 Mar 30;13:869754. doi: 10.3389/fphar.2022.869754. eCollection 2022. PMID 35444542
- [Background] Stiller CA, Trama A, Serraino D, Rossi S, Navarro C, Chirlaque MD, Casali PG; RARECARE Working Group. Descriptive epidemiology of sarcomas in Europe: report from the RARECARE project. Eur J Cancer. 2013 Feb;49(3):684-95. doi: 10.1016/j.ejca.2012.09.011. Epub 2012 Oct 15. PMID 23079473
- [Background] Rizvi NA, Hellmann MD, Brahmer JR, Juergens RA, Borghaei H, Gettinger S, Chow LQ, Gerber DE, Laurie SA, Goldman JW, Shepherd FA, Chen AC, Shen Y, Nathan FE, Harbison CT, Antonia S. Nivolumab in Combination With Platinum-Based Doublet Chemotherapy for First-Line Treatment of Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Sep 1;34(25):2969-79. doi: 10.1200/JCO.2016.66.9861. Epub 2016 Jun 27. PMID 27354481
- [Background] Sok M, Sentjurc M, Schara M, Stare J, Rott T. Cell membrane fluidity and prognosis of lung cancer. Ann Thorac Surg. 2002 May;73(5):1567-71. doi: 10.1016/s0003-4975(02)03458-6. PMID 12022551
- [Background] Subbiah V, Hess KR, Khawaja MR, Wagner MJ, Tang C, Naing A, Fu S, Janku F, Piha-Paul S, Tsimberidou AM, Herzog CE, Ludwig JA, Patel S, Ravi V, Benjamin RS, Meric-Bernstam F, Hong DS. Evaluation of Novel Targeted Therapies in Aggressive Biology Sarcoma Patients after progression from US FDA approved Therapies. Sci Rep. 2016 Oct 17;6:35448. doi: 10.1038/srep35448. PMID 27748430
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295